CLINICAL TRIAL: NCT03537079
Title: Hypoxic Conditioning Combined With Exercise Training in Heart Failure Patient: a Randomised, Controled, Single Blind Study
Brief Title: Hypoxic Conditioning in Heart Failure
Acronym: hypoxheart
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 38RC17.347
Record Dates: First submitted 2018-04-26; First posted 2018-05-25 (Actual); Last update posted 2020-03-25 (Actual); Status verified 2020-03

CONDITIONS: Heart Failure, Systolic
Keywords: hypoxia; exercise training; heart failure; cardiac remodeling
MeSH Terms: conditions — Heart Failure, Systolic; Hypoxia; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Masking Description: this is a single blind study patients don't know if they are breathing normal air (normoxia) or hypoxic air (hypoxia).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- normoxia conditioning (Placebo Comparator): exercise training in normoxia and rest conditioning in normoxia
  Interventions: Other: hypoxia air
- exercise hypoxia (Active Comparator): exercise training in hypoxia and rest conditioning in normoxia
  Interventions: Other: hypoxia air
- rest hypoxia (Active Comparator): exercise training in normoxia and rest conditioning in hypoxia
  Interventions: Other: hypoxia air

INTERVENTIONS:
Other: hypoxia air — Normobaric hypoxia is generated by adding azote in normal air to decrease the oxygen availability.

SUMMARY:
Heart failure impairs quality of life and exercise capacity, despite an optimal medical therapy. Alternative methods, like hypoxic conditioning coupled to exercise training, must be explored and describe

DETAILED DESCRIPTION:
All heart failure patients will have a session of 45' of bicycle exercise training (in normoxia or hypoxia) AND a one hour rest session (in normoxia or hypoxia).

Exercise training sessions will consist in a continue bicycle exercise test at 70 to 80 % of the maximal heart rate, while breathing (single blind) normoxia or hypoxia gaz.

Rest conditioning consist in a one hour of rest, while breathing (single blind) normoxia or hypoxia gaz.

For hypoxia sessions, the oxygen saturation target will be fo 85-90 % for the 4 first weeks and 80-85 % for the last 4 weeks.

Three arms :

* exercise training in NORMOXIA and rest conditioning in NORMOXIA
* exercise training in HYPOXIA and rest conditioning in NORMOXIA
* exercise training in NORMOXIA and rest conditioning in HYPOXIA

ELIGIBILITY:
Inclusion Criteria:

* patient available for exercise training
* stable heart failure state I-II New York Heart Association (NYHA) with altered ejection fraction (EF ≤ 40 %)
* signed informed consent

Exclusion Criteria:

* unstable ischemic cardiopathy
* right ventricle dysfunction
* uncontrolled arrythmias
* rest elevated in pulmonary artery pressure (≥ 45 mmHg)
* migraine
* high altitude trip above 2500 m high during study period
* impossibility to realise a maximal bicycle exercise test

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Estimated)
Dates: Start 2020-05 (Estimated); Primary Completion 2021-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
maximal oxygen uptake in ml/min/kg | after 8 weeks of training and conditioning
  The maximal exercise capacity will be assessed by an incremental maximal bicycle exercise test

SECONDARY OUTCOMES:
End diastolic left ventricle diameter in mm | After 8 weeks of training and conditioning
  In parasternal long axe, the end diastolic left ventricle diameter
systolic left ventricle ejection fraction in % | After 8 weeks of training and conditioning
  the systolic left ventricle ejection fraction will be assessed by Simpson's method in 4 and 2 cavity views
flow mediated dilatation (FMD) in % | After 8 weeks of training and conditioning
  The rest FMD will be assessed by echocardiography by using the % of variation of the brachial artery diameter 10 minutes after occlusion.
systolic and diastolic blood pressure control in mmHg | After 8 weeks of training and conditioning
  24 hours ambulatory blood pressure monitoring

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital, Grenoble, France